CLINICAL TRIAL: NCT05003180
Title: SunBurst (StUdy oN Burst Fractures) - a National, Multicenter, Register-based, Randomized Controlled Trial on Thoracolumbar Burst Fractures
Brief Title: StUdy oN Burst Fractures (SunBurst)
Acronym: SunBurst
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Uppsala University Hospital (Other); University Hospital, Umeå (Other); University Hospital, Linkoeping (Other); Skane University Hospital (Other); Region Örebro County (Other); Stockholm South General Hospital (Other); Karolinska University Hospital (Other); Oslo University Hospital (Other); Haukeland University Hospital (Other); Helse Stavanger HF (Other Government); University Hospital, Akershus (Other); Kalmar County Hospital (Other); Ryhov County Hospital (Other); Halmstad County Hospital (Other); Centrallasarettet Västerås (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Paul Gerdhem, MD, PhD, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB-PG-PF-OW-SM-2021-SunBurst; 2020-00493 (Other Grant/Funding Number: The Swedish Research Council); No grant number (Other Grant/Funding Number: The Swedish Society of Spinal Surgeons); RV-1010099, RV-1030408 (Other Grant/Funding Number: ALF medel Region Västerbotten)
Record Dates: First submitted 2021-06-20; First posted 2021-08-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Thoracolumbar Burst Fracture
Keywords: Thoracolumbar spine; Burst fractures; Thoracic or lumbar vertebrae; Register-based; Randomized controlled trial; Conservative treatment; Surgical treatment; Non-surgical treatment

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Subjects are identified through spine services at hospitals throughout Sweden and Norway. The subjects are screened for eligibility. Subjects are randomized in a 1:1 ratio to surgical or non-surgical treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical (Active Comparator): Surgical stabilization. Brace treatment will not be used postoperative. Early ambulation after surgery is encouraged. Surgery is to be performed within 2 weeks from the injury. The choice of supplier and brand of implants are based on the preference of each participating center.
  Physiotherapy and other measures of rehabilitation are prescribed on an individual basis.
  Interventions: Procedure: Surgical stabilization
- Non-surgical treatment (No Intervention): No surgical stabilization is performed. Early ambulation after treatment randomization is encouraged. Brace treatment is not required, but a standard three-point hyperextension brace may be offered up to 3 months for pain relief. The choice of supplier and brand of brace are based on the preference of each participating center. The brace will only be used upon mobilization. Brace use will be estimated by the patient at the 3-4 months follow-up.
  Physiotherapy and other measures of rehabilitation are prescribed on an individual basis.

INTERVENTIONS:
Procedure: Surgical stabilization — The surgical stabilization can be either open or minimally invasive. The recommended procedure is posterior fixation with pedicle screws and rods. Both short and long segment fixation are allowed in the study. It is up to the treating surgeon to decide on fusion or decompression. If feasible, pedicle screws are inserted in the fractured vertebra.
  Arms: Surgical

SUMMARY:
Thoracolumbar (TL) burst fractures are seen in all ages and usually associated with high-energy trauma. Treatment include both surgical and non-surgical options. In cases without neurological deficit or definite rupture of the posterior ligament complex (PLC) both surgical treatment and non-surgical treatment are considered standard of care. This study aims to compare outcome between surgical and non-surgical in patients with a single level TL burst fracture (AO A3/4) in a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The study is an international, multicenter, randomized controlled trial. 202 patients with a single level TL burst fracture will be enrolled in the study. They will be randomized 1:1 to either surgery or non-surgical treatment. The study is pragmatical in its approach, i.e., the treating physician can decide on details of the surgical treatment as well as details of the non-surgical treatment. In non-surgically treated patients brace treatment is not required, but a hyperextension brace may be offered. The subjects will be followed with patient reported outcomes, clinical assessments, and radiological assessments. Data will be collected from questionnaires, patient files or national registers to compare sick leave, medical complications, pharmaceutical prescriptions and overall costs for each treatment.

ELIGIBILITY:
Inclusion Criteria:

* A single level thoracolumbar (Th10-L3) burst fracture, A3 or A4, according to the AO Spine classification
* Aged 18-66 years
* Informed consent
* Acute injury with diagnosis and treatment within 2 weeks
* May have minor fractures in adjacent vertebras if these fractures in themselves would not have resulted in any treatment
* May have a single nerve root injury

Exclusion Criteria:

* Unable to consent, no consent given or not informed
* Neurological injury involving more than a single level root, i.e., spinal cord and/or cauda equina injury
* Definite rupture of the posterior tension band (through bony and/or ligamentous structures) verified on MRI
* Patients with ankylosing spinal disorders spanning the fracture area
* Prior spinal surgeries within the fractured area
* Open vertebral fracture
* Additional injury which would impair early ambulation, e.g., long bone fractures, severe head injury, long-lasting intensive care
* Patients not deemed suitable due to severe co-morbidities. (E.g., established osteoporosis that would impair the possibility to maintain integrity of spinal implants, pathological fractures, severe cardiac or pulmonary compromise, or other systemic disease that would result in such high anesthesiologic risk that surgery would not be attempted.)
* Patients already included in the study cannot be randomized again if they get an additional spine fracture

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Group difference in Oswestry Disability Index (ODI) 1 year after the fracture. | At 1 year after the fracture
  ODI is a patient-reported outcome measure for spinal disorders. It consists of 10 questions related to back specific disabilities such as pain, personal care, walking and sitting ability, lifting capacity and social life.

SECONDARY OUTCOMES:
Categories of Oswestry Disability Index (ODI) 1 year after the fracture | At 1 year after the fracture
  ODI is a patient-reported outcome measure for spinal disorders. It consists of 10 questions related to back specific disabilities such as pain, personal care, walking and sitting ability, lifting capacity and social life and can be summed to an ODI 0-100 score. Participants will be dichotomised based on their ODI score (0-20 vs. 21-100). We will compare the proportions between groups. This is a secondary analysis of the primary outcome.
Group difference in Oswestry Disability Index (ODI) 1 year after the fracture, adjusted. | At 1 year after the fracture.
  ODI is a patient-reported outcome measure for spinal disorders. It consists of 10 questions related to back specific disabilities such as pain, personal care, walking and sitting ability, lifting capacity and social life. The between-group difference in ODI at 1 year will be compared using linear regression adjusting for age, sex and fracture type (A3 vs A4). This will be part of a sensitivity analysis of the primary outcome.
Group difference in Oswestry Disability Index (ODI) first item (pain) 1 year after the fracture | At 1 year after the fracture
  ODI is a patient-reported outcome measure for spinal disorders. It consists of 10 questions related to back specific disabilities such as pain, personal care, walking and sitting ability, lifting capacity and social life. The first item pain will be separately analysed as part of a sensitivity analysis of the primary outcome.
Group difference in Oswestry Disability Index (ODI) 3-4 months after the fracture | At 3-4 months after the fracture.
  ODI is a patient-reported outcome measure for spinal disorders. It consists of 10 questions related to back specific disabilities such as pain, personal care, walking and sitting ability, lifting capacity and social life.
Categories of Oswestry Disability Index (ODI) 3-4 months after the fracture | At 3-4 months after the fracture
  ODI is a patient-reported outcome measure for spinal disorders. It consists of 10 questions related to back specific disabilities such as pain, personal care, walking and sitting ability, lifting capacity and social life and can be summed to an ODI 0-100 score. Participants will be dichotomised based on their ODI score (0-20 vs. 21-100). We will compare the proportions between groups.
Group difference in Oswestry Disability Index (ODI) first item (pain) 3-4 months after the fracture | At 3-4 months after the fracture
  ODI is a patient-reported outcome measure for spinal disorders. It consists of 10 questions related to back specific disabilities such as pain, personal care, walking and sitting ability, lifting capacity and social life.
Change in Oswestry Disability Index (ODI) from baseline (prior injury) to 3-4 months after the fracture | At enrollment to 3-4 months after the fracture.
  Change in ODI between groups.
Change in Oswestry Disability Index (ODI) from baseline (prior injury) to 1 year after the fracture | At enrollment to 1 year after the fracture.
  Change in ODI between groups.
Group difference in Short Musculoskeletal Function Assessment (SMFA) at 3-4 months | At 3-4 months after the fracture.
  SMFA is a patient-reported outcome measure for a broad range of musculoskeletal disorders consisting of a total of 46 questions. 34 questions measure the patient's dysfunction and 12 questions measure how bothered the patients are by their symptoms.
Group difference in Short Musculoskeletal Function Assessment (SMFA) at 1 year | At 1 year after the fracture.
  SMFA is a patient-reported outcome measure for a broad range of musculoskeletal disorders consisting of a total of 46 questions. 34 questions measure the patient's dysfunction and 12 questions measure how bothered the patients are by their symptoms.
Change in Short Musculoskeletal Function Assessment (SMFA) from baseline (prior injury) to 3-4 months after the fracture | At enrollment to 3-4 months after the fracture.
  Change in SMFA between groups.
Change in Short Musculoskeletal Function Assessment (SMFA) from the time of the fracture to 1 year after the fracture | At enrollment to 1 year after the fracture.
  Change in SMFA between groups.
Group difference in EQ-5D-5L at 3-4 months | At 3-4 months after the fracture.
  EQ-5D-5L is a standardized quality of life instrument developed by the EuroQol group. It consists of 5 dimensions measuring mobility, personal care, usual activities, pain/discomfort and anxiety/depression with 5 levels for each dimension (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, 5=extreme problems). It also has a visual analog scale (EQ VAS) from 0 (worst possible health) to 100 (best possible health) to measure how the subjects consider their own health.
Group difference in EQ-5D-5L at 1 year | At 1 year after the fracture.
  EQ-5D-5L is a standardized quality of life instrument developed by the EuroQol group. It consists of 5 dimensions measuring mobility, personal care, usual activities, pain/discomfort and anxiety/depression with 5 levels for each dimension (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, 5=extreme problems). It also has a visual analog scale (EQ VAS) from 0 (worst possible health) to 100 (best possible health) to measure how the subjects consider their own health.
Change in EQ-5D-5L from baseline (prior injury) to 3-4 months after the fracture | At enrollment to 3-4 months after the fracture.
  Change in EQ-5D-5L between groups.
Change in EQ-5D-5L from baseline (prior injury) to 1 year after the fracture | At enrollment to 1 year after the fracture.
  Change in EQ-5D-5L between groups.
Group difference in radiographic fracture pattern- standing radiograph | At 1 year after the fracture.
  The patients will do a standing, whole spine radiograph. The degree of fracture compression, local and global kyphosis will be registered.
Group difference in radiographic pattern- supine computed tomography at 1 year | At 1 year after the fracture.
  The patients will do a computed tomography (CT) 1 year after the fracture. The degree of fracture compression, local and global kyphosis and adjacent segment degeneration will be compared.
Group difference in radiographic pattern- supine computed tomography at 3-4 months | At 3-4 months after the fracture.
  The patients will do a computed tomography (CT) at 3-4 months after the fracture. The degree of fracture compression, local and global kyphosis and adjacent segment degeneration will be compared.
Change in radiographic pattern- supine computed tomography - from the time of fracture to 3-4 months | From the time of fracture to 3-4 months after the fracture.
  The patients will do a computed tomography (CT). The degree of fracture compression, local and global kyphosis and adjacent segment degeneration will be registered. Group comparisons of radiological changes will be performed.
Change in radiographic pattern- supine computed tomography - from 3-4 months to 1 year from the fracture | From 3-4 months after the fracture to 1 year after the fracture.
  The patients will do a computed tomography (CT). The degree of fracture compression, local and global kyphosis and adjacent segment degeneration will be registered. Group comparisons of radiological changes will be performed.
Change in radiographic pattern- supine computed tomography - from the time of fracture to 1 year | From the time of fracture to 1 year after the fracture.
  The patients will do a computed tomography (CT). The degree of fracture compression, local and global kyphosis and adjacent segment degeneration will be registered. Group comparisons of radiological changes will be performed.
Magnetic resonance imaging (MRI) at 1 year | At 1 year after the fracture.
  The patients will do a magnetic resonance imaging (MRI). The degree of fracture compression, local and global kyphosis, adjacent segment degeneration and extent of any soft tissue injuries will be registered. Group comparisons of MRI changes will be performed.
Imaging in correlation to patient reported outcome measures at 3-4 months from the fracture | At 3-4 months from the fracture.
  The degree of fracture compression, local and global kyphosis, adjacent segment degeneration and extent of any soft tissue injuries registered on computed tomography (CT) will be compared to patient reported outcome measures at 3 to 4 months.
Imaging in correlation to patient reported outcome measures at 1 year from the fracture | At 1 year after the fracture.
  The degree of fracture compression, local and global kyphosis, adjacent segment degeneration and extent of any soft tissue injuries registered on X-ray, CT and MRI will be compared to patient reported outcome measures at 1 year.
Adverse events | 1 year after last subject recruitment
  Adverse events will be collected from medical records and patient-reported questionnaires, the National Patient Register administered by the National Board of Health and Welfare and the Swedish Fracture register in Sweden. For participants treated in Norway, corresponding data will be collected from medical records and patient-reported questionnaires. The number of adverse events will be compared between the study groups.
Drug prescription/consumption | 1 year after last subject recruitment
  Data on prescribed analgesics and antibiotics will be obtained from the Swedish Prescribed Drug Register administered by the National Board of Health and Welfare. Prescription data will be analyzed as dichotomous variables (yes/no) for predefined time intervals: 0-4 months and 4-12 months following injury.
  For participants treated in Norway, corresponding information will be collected through review of medical records and patient-reported questionnaires.
Sick leave | 1 year after inclusion
  Data from the Swedish Social Insurance Agency / Statistics Sweden will be collected to compare sick leave and loss of income due to the fracture. Data will be stratified based on the presence or absence of sick leave before the fracture event. Data on total time on sick leave as well as the diagnosis used for sick leave will be collected. In Norway similar data will be collected from the patient files and questionnaires.
Individual cost from the time of fracture to 3-4 months | From the time of fracture to 3-4 months after the fracture.
  The number of outpatient and telephone contacts (physician, nurse, physiotherapist) and salary losses the fracture and treatment have resulted in will be collected from patient files and official health registries and compared between the groups.
Individual cost from the time of fracture to 1 year | From the time of fracture to 1 year after the fracture.
  The number of outpatient and telephone contacts (physician, nurse, physiotherapist) and salary losses the fracture and treatment have resulted in will be collected from patient files and official health registries and compared between the groups.
Incremental cost-effectiveness ratio | 1 year after last subject recruitment
  Quality-adjusted life years (QALYs) will be calculated for each group as measured by EQ-5D-5L. Combining cost and QALY yields the incremental cost-effectiveness ratio (ICER) of the surgical intervention as compared to non-surgical care.
Mortality at 1 year | 1 year after last subject recruitment
  Mortality, including the cause of death, will be collected from the National Board of Health and Welfare Cause of Death Register. In Norway data will be collected from official registries.
Mortality at 5 year | 5 years after last subject recruitment
  Mortality, including the cause of death, will be collected from the National Board of Health and Welfare Cause of Death Register. In Norway data will be collected from official registries.
Mortality at 10 years | 10 years after last subject recruitment
  Mortality, including the cause of death, will be collected from the National Board of Health and Welfare Cause of Death Register. In Norway data will be collected from official registries.
Oswestry Disability index (ODI) at 5 years | At 5 years after the fracture.
  ODI are planned to be collected at 5 years.
Oswestry Disability index (ODI) at 10 years | At 10 years after the fracture.
  ODI are planned to be collected at 10 years.
Short Musculoskeletal Function Assessment (SMFA) at 5 years | At 5 years after the fracture.
  SMFA are planned to be collected after 5 years.
Short Musculoskeletal Function Assessment (SMFA) at 10 years | At10 years after the fracture.
  SMFA are planned to be collected after 10 years.
EQ-5D-5L at 5 years | At 5 years after the fracture.
  EQ-5D-5L are planned to be collected after 5 years.
EQ-5D-5L at 10 years | At10 years after the fracture.
  EQ-5D-5L are planned to be collected after 10 years.
Sick leave at 5 years | At 5 years after the fracture.
  Long-term data on sick leave are to be collected from the Social Insurance Agency at 5 years to compare difference in long-term sick leave between study groups. In Norway similar data will be collected from patient files and questionnaires.
Sick leave at 10 years | At 10 years after the fracture.
  Long-term data on sick leave are to be collected from the Social Insurance Agency at 10 years to compare difference in long-term sick leave between study groups. In Norway similar data will be collected from patient files and questionnaires.
Social cost at 5 years | At 5 years after the fracture.
  Analysis of the long-term social cost will be calculated for each treatment by collecting data on cost from sick leave from the Social Insurance Agency, estimated cost from health care visits collected from the National Patient Register and estimated cost on pharmaceutical prescriptions from the Prescribed Drug Register at 5 years. In Norway similar data will be collected from patient files and questionnaires.
Social cost at 10 years | At 10 years after the fracture.
  Analysis of the long-term social cost will be calculated for each treatment by collecting data on cost from sick leave from the Social Insurance Agency, estimated cost from health care visits collected from the National Patient Register and estimated cost on pharmaceutical prescriptions from the Prescribed Drug Register at 10 years. In Norway similar data will be collected from patient files and questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gerdhem, MD, PhD, Principal Investigator — Uppsala University, Uppsala University Hospital and Karolinska Institutet; Filip Dolatowski, MD, PhD, Study Director — Oslo University Hospital
Locations (17):
- Norway (5):
  - Oslo University Hospital, Oslo, Oslo County
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - St. Olavs Hospital, Trondheim
- Sweden (12):
  - Sahlgrenska University Hospital, Gothenburg, Gothenburg
  - Linköping University Hospital, Linköping, Linköping
  - Skåne University Hospital, Malmo, Malmö
  - Stockholm South General Hospital, Stockholm, Stockholm County
  - University Hospital of Umeå, Umeå, Umeå
  - Uppsala University Hospital, Uppsala, Uppsala County
  - Halmstad Hospital, Halmstad
  - Ryhov Hospital, Jönköping
  - Kalmar Hospital, Kalmar
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Central Hospital of Västerås, Västerås

IPD SHARING:
Plan to Share IPD: Yes
IPD underlying the results reported in publications will be shared in a pseudonymized form with external researchers only if required approvals are in place. Data can only be made available subject to approval by the Swedish ethical authority, appropriate data sharing agreements, and compliance with applicable data protection legislation.
Supporting Information: Study Protocol, SAP
Time Frame: IPD:
  Beginning after publication of the primary study results.
  Supporting information:
  Study protocol: is attached. Statistical analysis plan: Is attached
Access Criteria: Access to pseudonymized individual participant data will only be granted following approval by the Swedish ethical authority and completion of appropriate data sharing agreements. The investigators in charge will administer access in accordance with applicable data protection legislation.

REFERENCES:
- [Background] Rajasekaran S, Kanna RM, Shetty AP. Management of thoracolumbar spine trauma: An overview. Indian J Orthop. 2015 Jan-Feb;49(1):72-82. doi: 10.4103/0019-5413.143914. PMID 25593358
- [Background] Schouten R, Lewkonia P, Noonan VK, Dvorak MF, Fisher CG. Expectations of recovery and functional outcomes following thoracolumbar trauma: an evidence-based medicine process to determine what surgeons should be telling their patients. J Neurosurg Spine. 2015 Jan;22(1):101-11. doi: 10.3171/2014.9.SPINE13849. PMID 25396259
- [Background] Gnanenthiran SR, Adie S, Harris IA. Nonoperative versus operative treatment for thoracolumbar burst fractures without neurologic deficit: a meta-analysis. Clin Orthop Relat Res. 2012 Feb;470(2):567-77. doi: 10.1007/s11999-011-2157-7. Epub 2011 Nov 5. PMID 22057820
- [Background] Vaccaro AR, Schroeder GD, Kepler CK, Cumhur Oner F, Vialle LR, Kandziora F, Koerner JD, Kurd MF, Reinhold M, Schnake KJ, Chapman J, Aarabi B, Fehlings MG, Dvorak MF. The surgical algorithm for the AOSpine thoracolumbar spine injury classification system. Eur Spine J. 2016 Apr;25(4):1087-94. doi: 10.1007/s00586-015-3982-2. Epub 2015 May 8. PMID 25953527
- [Background] Oner C, Rajasekaran S, Chapman JR, Fehlings MG, Vaccaro AR, Schroeder GD, Sadiqi S, Harrop J. Spine Trauma-What Are the Current Controversies? J Orthop Trauma. 2017 Sep;31 Suppl 4:S1-S6. doi: 10.1097/BOT.0000000000000950. PMID 28816869
- [Background] Yi L, Jingping B, Gele J, Baoleri X, Taixiang W. Operative versus non-operative treatment for thoracolumbar burst fractures without neurological deficit. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD005079. doi: 10.1002/14651858.CD005079.pub2. PMID 17054237
- [Background] van der Roer N, de Lange ES, Bakker FC, de Vet HC, van Tulder MW. Management of traumatic thoracolumbar fractures: a systematic review of the literature. Eur Spine J. 2005 Aug;14(6):527-34. doi: 10.1007/s00586-004-0847-5. Epub 2005 Feb 3. PMID 15690209
- [Background] Dai LY, Jiang SD, Wang XY, Jiang LS. A review of the management of thoracolumbar burst fractures. Surg Neurol. 2007 Mar;67(3):221-31; discussion 231. doi: 10.1016/j.surneu.2006.08.081. PMID 17320622
- [Background] Rometsch E, Spruit M, Hartl R, McGuire RA, Gallo-Kopf BS, Kalampoki V, Kandziora F. Does Operative or Nonoperative Treatment Achieve Better Results in A3 and A4 Spinal Fractures Without Neurological Deficit?: Systematic Literature Review With Meta-Analysis. Global Spine J. 2017 Jun;7(4):350-372. doi: 10.1177/2192568217699202. Epub 2017 Jul 7. PMID 28815163
- [Background] Abudou M, Chen X, Kong X, Wu T. Surgical versus non-surgical treatment for thoracolumbar burst fractures without neurological deficit. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD005079. doi: 10.1002/14651858.CD005079.pub3. PMID 23740669
- [Background] Ghobrial GM, Maulucci CM, Maltenfort M, Dalyai RT, Vaccaro AR, Fehlings MG, Street J, Arnold PM, Harrop JS. Operative and nonoperative adverse events in the management of traumatic fractures of the thoracolumbar spine: a systematic review. Neurosurg Focus. 2014;37(1):E8. doi: 10.3171/2014.4.FOCUS1467. PMID 24981907
- [Background] Wallace N, McHugh M, Patel R, Aleem IS. Effects of Bracing on Clinical and Radiographic Outcomes Following Thoracolumbar Burst Fractures in Neurologically Intact Patients: A Meta-Analysis of Randomized Controlled Trials. JBJS Rev. 2019 Sep;7(9):e9. doi: 10.2106/JBJS.RVW.19.00006. PMID 31567716
- [Background] Emilsson L, Lindahl B, Koster M, Lambe M, Ludvigsson JF. Review of 103 Swedish Healthcare Quality Registries. J Intern Med. 2015 Jan;277(1):94-136. doi: 10.1111/joim.12303. Epub 2014 Sep 27. PMID 25174800
- [Background] Wennergren D, Moller M. Implementation of the Swedish Fracture Register. Unfallchirurg. 2018 Dec;121(12):949-955. doi: 10.1007/s00113-018-0538-z. PMID 30178109
- [Background] Wolf O, Mukka S, Notini M, Moller M, Hailer NP; DUALITY GROUP. Study protocol: The DUALITY trial-a register-based, randomized controlled trial to investigate dual mobility cups in hip fracture patients. Acta Orthop. 2020 Oct;91(5):506-513. doi: 10.1080/17453674.2020.1780059. Epub 2020 Jun 22. PMID 32567472
- [Background] Wolf O, Sjoholm P, Hailer NP, Moller M, Mukka S. Study protocol: HipSTHeR - a register-based randomised controlled trial - hip screws or (total) hip replacement for undisplaced femoral neck fractures in older patients. BMC Geriatr. 2020 Jan 21;20(1):19. doi: 10.1186/s12877-020-1418-2. PMID 31964340
- [Background] Vaccaro AR, Oner C, Kepler CK, Dvorak M, Schnake K, Bellabarba C, Reinhold M, Aarabi B, Kandziora F, Chapman J, Shanmuganathan R, Fehlings M, Vialle L; AOSpine Spinal Cord Injury & Trauma Knowledge Forum. AOSpine thoracolumbar spine injury classification system: fracture description, neurological status, and key modifiers. Spine (Phila Pa 1976). 2013 Nov 1;38(23):2028-37. doi: 10.1097/BRS.0b013e3182a8a381. PMID 23970107
- [Background] Reinhold M, Audige L, Schnake KJ, Bellabarba C, Dai LY, Oner FC. AO spine injury classification system: a revision proposal for the thoracic and lumbar spine. Eur Spine J. 2013 Oct;22(10):2184-201. doi: 10.1007/s00586-013-2738-0. Epub 2013 Mar 19. PMID 23508335
- [Background] James S, Rao SV, Granger CB. Registry-based randomized clinical trials--a new clinical trial paradigm. Nat Rev Cardiol. 2015 May;12(5):312-6. doi: 10.1038/nrcardio.2015.33. Epub 2015 Mar 17. PMID 25781411
- [Background] Ni WF, Huang YX, Chi YL, Xu HZ, Lin Y, Wang XY, Huang QS, Mao FM. Percutaneous pedicle screw fixation for neurologic intact thoracolumbar burst fractures. J Spinal Disord Tech. 2010 Dec;23(8):530-7. doi: 10.1097/BSD.0b013e3181c72d4c. PMID 21131801
- [Background] Chi JH, Eichholz KM, Anderson PA, Arnold PM, Dailey AT, Dhall SS, Harrop JS, Hoh DJ, Qureshi S, Rabb CH, Raksin PB, Kaiser MG, O'Toole JE. Congress of Neurological Surgeons Systematic Review and Evidence-Based Guidelines on the Evaluation and Treatment of Patients With Thoracolumbar Spine Trauma: Novel Surgical Strategies. Neurosurgery. 2019 Jan 1;84(1):E59-E62. doi: 10.1093/neuros/nyy364. PMID 30299485
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Vianin M. Psychometric properties and clinical usefulness of the Oswestry Disability Index. J Chiropr Med. 2008 Dec;7(4):161-3. doi: 10.1016/j.jcm.2008.07.001. PMID 19646379
- [Background] Ponzer S, Skoog A, Bergstrom G. The Short Musculoskeletal Function Assessment Questionnaire (SMFA): cross-cultural adaptation, validity, reliability and responsiveness of the Swedish SMFA (SMFA-Swe). Acta Orthop Scand. 2003 Dec;74(6):756-63. doi: 10.1080/00016470310018324. PMID 14763711
- [Background] Burstrom K, Teni FS, Gerdtham UG, Leidl R, Helgesson G, Rolfson O, Henriksson M. Experience-Based Swedish TTO and VAS Value Sets for EQ-5D-5L Health States. Pharmacoeconomics. 2020 Aug;38(8):839-856. doi: 10.1007/s40273-020-00905-7. PMID 32307663
- [Background] Hagg O, Fritzell P, Nordwall A; Swedish Lumbar Spine Study Group. The clinical importance of changes in outcome scores after treatment for chronic low back pain. Eur Spine J. 2003 Feb;12(1):12-20. doi: 10.1007/s00586-002-0464-0. Epub 2002 Oct 24. PMID 12592542
- [Background] Copay AG, Glassman SD, Subach BR, Berven S, Schuler TC, Carreon LY. Minimum clinically important difference in lumbar spine surgery patients: a choice of methods using the Oswestry Disability Index, Medical Outcomes Study questionnaire Short Form 36, and pain scales. Spine J. 2008 Nov-Dec;8(6):968-74. doi: 10.1016/j.spinee.2007.11.006. Epub 2008 Jan 16. PMID 18201937
- [Background] Jonas WB, Crawford C, Colloca L, Kaptchuk TJ, Moseley B, Miller FG, Kriston L, Linde K, Meissner K. To what extent are surgery and invasive procedures effective beyond a placebo response? A systematic review with meta-analysis of randomised, sham controlled trials. BMJ Open. 2015 Dec 11;5(12):e009655. doi: 10.1136/bmjopen-2015-009655. PMID 26656986
- [Derived] Blixt S, Mukka S, Forsth P, Westin O, Gerdhem P; SunBurst study group. Study protocol: The SunBurst trial-a register-based, randomized controlled trial on thoracolumbar burst fractures. Acta Orthop. 2022 Jan 24;93:256-263. doi: 10.2340/17453674.2022.1614. PMID 35175357
- See also: Information on the National Board of Health and Welfare,The National Patient Register. — https://www.socialstyrelsen.se/statistik-och-data/register/patientregistret/
- See also: Information on the National Board of Health and Welfare, The Swedish Prescribed Drug Register. — https://www.socialstyrelsen.se/statistik-och-data/register/lakemedelsregistret/
- See also: Information in Swedish on the National Board of Health and Welfare, Cause of Death Register (Socialstyrelsen. Dödsorsaksregistret.) — https://www.socialstyrelsen.se/statistik-och-data/register/dodsorsaksregistret/